CLINICAL TRIAL: NCT03540355
Title: Phase III, National, Multicenter, Randomized, Double-blind Clinical Trial, to Evaluate the Efficacy and Safety of Cipros 20 Association on the Dyslipidemia Treatment
Brief Title: Efficacy and Safety of Cipros 20 Association on Dyslipidemia Treatment
Acronym: CIPROS20
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0717
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cipros 20 (Experimental): The study is double-masked, the patient will take 2 tablets, as follow:
  1 tablet Cipros 20 association; and
  1 tablet crestor placebo. Oral, once a day
  Interventions: Drug: Cipros 20 association
- Crestor (Active Comparator): The study is double-masked, the patient will take 2 tablets, as follow:
  1 tablet Crestor 20 mg; and
  1 tablet cipros association placebo. Oral, once a day
  Interventions: Drug: Crestor 20 mg

INTERVENTIONS:
Drug: Cipros 20 association — oral, once a day
  Other Names: EMS Association
  Arms: Cipros 20
Drug: Crestor 20 mg — Oral, once a day
  Other Names: Rosuvastatin 20 mg
  Arms: Crestor

SUMMARY:
The purpose of this study is to evaluate the efficacy of Cipros 20 association in the treatment of dyslipidemia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes, aged 18 years or more;
* Participants with the diagnosed of dyslipidemia and with high or very high cardiovascular risk, according to the Brazillian Guidelines on Dyslipidemia and Prevention of Atherosclerosis;
* Signed consent.

Exclusion Criteria:

* Using medications that may interfere with the metabolism or serum levels of triglycerides;
* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Presence of concomitant cardiovascular disease, renal failure and hepatic failure;
* Decompensated diabetes;
* Current smoking;
* History hypersensitivity to the active ingredients used in the study;
* Pregnancy or risk of pregnancy and lactating patients;
* History of alcohol abuse or illicit drug use;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Reduction of serum triglyceride levels | 12 weeks vs baseline
  The reduction of triglyceride levels will be measured through the difference of values in the first visit and last visit.
Reduction of serum LDL-c | 12 weeks vs baseline
  The reduction of serum-LDL-c will be measured through the difference of values in the first and last visit.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided